CLINICAL TRIAL: NCT02667028
Title: Retrospective Evaluation of Prognosis of Pci Patients Using Network Data in SHengjing Hospital of China Medical University
Brief Title: Retrospective Evaluation of Prognosis of Pci Patients Using Network Data in SHengjing Hospital
Acronym: R-PUSH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, YU Tong-tong, attending physician, Shengjing Hospital
Other Study IDs: 2016PS04K01
Record Dates: First submitted 2016-01-19; First posted 2016-01-28 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients receiving PCI: patients receiving percutaneous coronary intervention(PCI)
  Interventions: Procedure: PCI

INTERVENTIONS:
Procedure: PCI — percutaneous coronary intervention

SUMMARY:
Coronary heart disease (CHD) has a serious health threaten to population. PCI is a well-proved measure in CHD management. However, the knowledge about the real-life PCI use and how evidence-based therapies in routine clinical practice is limited. In a large-scale hospital in Northeast China, the investigators will examine various factors of 3007 consecutive PCI inpatient cases from January 1, 2010 to October 31, 2014. The medical records will be reviewed and abstracted to evaluate the clinical treatment pattern and outcomes. Basic data and innovative evidence will accelerate evidence-based clinical practice, and improve patients' outcomes in future finally.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is a major concern in public health in China. Relatively limited information is available about how evidence-based therapies are incorporated appropriately into routine clinical practice. In addition, little information is available about the practical and applied knowledge from large unselected population and is used to guide practice for quality improvement.

To investigate the treatment pattern and outcomes of PCI in a real-world clinical setting, 3007 consecutive PCI cases will be selected from January 1, 2010 to October 31, 2014, in a large-scale hospital in Northeast China.At first, the investigators identified all PCI patients from PACS (Picture Archiving and Communication Systems) of the interventional imaging data from January 1, 2010 to October 31, 2014 and assigned each case a unique study ID. Then, the investigators abstracted comprehensive clinical data and procedural data. Comprehensive clinical data came from electronic medical records, including patient demographic characteristics, past cardiac and noncardiac history, patient clinical characteristics on hospital admission, laboratory measurements, procedure-related complications and use of cardiac medications during the index hospitalization and at discharge. CAG imaging will be reviewed by 2 cardiologists through PACS. Other Procedural data, including stent type, total stent length and so on, came from operation records of PCI cases finished by operators. The first clinical follow-up was assessed in October 2015 by direct hospital visits or phone interviews of patient's general practitioner/cardiologist, patient himself, or his family for all cases. A secondary clinical follow-up will be assessed individually if the three-year-follow-up of the patient was available. A third clinical follow-up will be assessed individually if the five-year-follow-up of the patient was available. All events were obtained from the patients' medical records. If these data were unavailable, status was ascertained by a telephone call to the patient's referring hospital physician. All events were adjudicated and classified by 2 cardiologists. By characterizing differences in patients' features, comparing the use of medications and procedures, and examining the outcomes, we'll define the gaps between clinical practice and guidelines to evaluated the treatment pattern and outcomes. New knowledge will be generated about PCI management to provide evidence for clinical guidelines, and to improve patients prognosis in future finally.

ELIGIBILITY:
Inclusion Criteria:

• Hospitalized patients undergoing a percutaneous coronary intervention (PCI) for coronary lesions.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients receiving PCI in department of Cardiology,Shengjing Hospital of China Medical University from January 1, 2010 to October 31, 2014
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2015-10; Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Major adverse cardiovascular events (MACE) | 5 years
  Composite of major adverse cardiovascular events (MACE) includes cardiac death, non-fatal AMI, coronary revascularization procedure.

SECONDARY OUTCOMES:
Percentage of Participants with all-cause death | 5 years
Percentage of Participants with cardiac death | 5 years
Percentage of Participants with non-fatal AMI | 5 years
Percentage of Participants with coronary revascularization | 5 years
  coronary revascularization includes any unplanned repeat PCI or surgical bypass of target or non-target vessels.
Percentage of Participants with stroke | 5 years
Percentage of Participants with Cardiac Re-admission | 5 years
  Cardiac Re-admission includes any re-admission because of aggravation of heart failure or angia.
Percentage of Participants with adherence to medications for secondary prevention | 5 years
  Taking the following medications for 6 or more days per week: aspirin, clopidogrel, ACEI/ARB, statin and beta-blockers
Number of Participants who quit smoking | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: tongtong yu, Doctor, Principal Investigator — Shengjing Hospital
Locations (1):
- Shengjing Hospital, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No
We will not share IPD to protect our data very well.